CLINICAL TRIAL: NCT06332547
Title: A Multicenter Prospective, Randomized Controlled Study of Different Transfusion Thresholds in Cardiac Valve Surgery
Brief Title: Transfusion in Cardiac Valve Surgery
Acronym: TICVS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TICVS
Record Dates: First submitted 2024-03-18; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Cardiac Surgery With Cardiopulmonary Bypass; Valve Heart Disease
Keywords: cardiac valve surgery; transfusion; transfusion threshold
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restrictive transfusion strategy (Active Comparator): Restrictive transfusion strategy: Blood transfusion triggers of Hb valve less than 6.0g/dL or Hct value less than 18% during CPB, Hb valve less than 7.0g/dL or Hct value less than 21% in ICU or general ward.
  Red blood cell transfusion will be given when Hct values fall below 18% or Hb fall below 6.0g/dL during CPB, 2 units RBC transfusion will be administered. In ICU or general ward after surgery, RBC transfusion will be given when Hct values fall below 21% or Hb fall below 7.0g/dL during CPB, 2 unit RBC transfusion will be administered. Following administration of the 2 units transfusion a repeat HCT or Hb is performed, if their values greater than threshold, no further transfusions will be administered, or will be received 2 units RBC again.
  Interventions: Other: Restrictive Transfusion Strategy
- Liberal Transfusion Strategy (Active Comparator): Liberal Transfusion Strategy: Blood transfusion triggers of Hb valve less than 8.0g/dL or Hct value less than 24% during CPB, Hb valve less than 10.0g/dL or Hct value less than 30% in ICU or general ward.
  Red blood cell transfusion will be given when Hct values fall below 24% or Hb fall below 8.0g/dL during CPB, 2 units RBC transfusion will be administered. In ICU or general ward after surgery, RBC transfusion will be given when Hct values fall below 30% or Hb fall below 10.0g/dL during CPB, 2 units RBC transfusion will be administered. Following administration of the 2 units transfusion a repeat HCT or Hb is performed, if their values greater than threshold, no further transfusions will be administered, or will be received 2 units RBC again.
  Interventions: Other: Liberal Transfusion Strategy

INTERVENTIONS:
Other: Restrictive Transfusion Strategy — Blood transfusion at HCT less than 21% or Hb less than 6.0g/dL during CPB, at HCT less than 21% or Hb less than 7.0g/dL in ICU or general ward after surgery
  Arms: Restrictive transfusion strategy
Other: Liberal Transfusion Strategy — Blood transfusion at HCT less than 24% or Hb less than 8.0g/dL during CPB, at HCT less than 30% or Hb less than 10.0g/dL in ICU or general ward after surgery
  Arms: Liberal Transfusion Strategy

SUMMARY:
This prospective, randomized controlled study is aimed to figure out suitable transfusion threshold in patients undergoing cardiac valve surgery under cardiopulmonary bypass(CPB). Patients are randomly assigned to restrictive and liberal transfusion group and receive blood transfusion during and after surgery. Compare primary and secondary outcomes of two groups.

DETAILED DESCRIPTION:
Patients are randomly assigned to restrictive-threshold group and liberal-threshold group before cardiac group. Patients are included in this research when their Hct meets 24% during CPB.

Arterial blood gas analysis will be done in 0.5h, 1.5h, 2.5h, 3.5h...after CPB start and 0.5h before CPB finish.

Arterial blood gas analysis will be done every 4h in intensive care unit(ICU) and everyday in general ward.

Restrictive-threshold group: The transfusion threshold is Hemoglobin(Hb) ≤ 6.0g/dL or Hct ≤ 18% during CPB; postoperative Hb ≤ 7.0g/dL or Hct ≤ 21% in ICU or general ward.

Liberal-threshold group: The transfusion threshold is Hb ≤ 8.0g/dL or Hct ≤ 24% during CPB; postoperative Hb ≤ 10.0g/dL or Hct ≤ 30% in ICU or general ward.

If the Hb or Hct fall below the threshold at any time, 2 unit of blood cells is administered as soon as possible. Test Hb or Hct again, if is under the threshold 2 unit blood cells will be given until reach the threshold.

ELIGIBILITY:
Inclusion Criteria:

* All cardiac valve surgical patients undergoing CPB, isolated valve procedures Informed consent obtained

Exclusion Criteria:

* Pregnant or maternal women Age less than 18 years or more than 80 years Undergo coronary artery bypass or large cardiac vessels procedure Emergencies Have been attended other researches Unable to receive blood for religious reasons Drug addict or malignant tumor patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
A composite of postoperative morbidity and mortality | Postoperative 6 months
  The composite components are postoperative mortality, infectious morbidity(wound infection, septicemia, or sepsis), ischemic event(myocardial infarction, stroke, renal infraction, bowel infraction )

SECONDARY OUTCOMES:
Rate of reoperation | Postoperative 6 months
Length of ICU Stays | From date of the end of operation until the date of discharging from ICU or date of death from any cause, whichever comes first, assessed up to 2 months.
Length of Postoperative Hospital Stay | From date of discharging from ICU until the date of discharging from hospital or date of death from any cause, whichever comes first, assessed up to 2 months.
Number of Blood Transfusion | From date of beginning of surgery until the date of discharging from hospital or date of death from any cause, whichever comes first, assessed up to 3 months.
Duration of mechanical ventilation | From date of the end of surgery until the date of discharging from ICU or date of death from any cause, whichever comes first, assessed up to 2 months.
Postoperative thoracic fluid volume in the first 24 hours | The first 24 hours after surgery
Number of participants with postoperative atrial fibrillation | Postoperative 6 months
Number of participants with new-onset renal failure with dialysis | Postoperative 6 months
Number of participants with acute kidney injury | Postoperative 6 months
Number of participants with delirium | Postoperative 6 months
Hospitalization expense | From date of being admitted to hospital until the date of discharging from hospital or date of death from any cause, whichever comes first, assessed up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Huang Huanlei, Phd, Principal Investigator — hhuanlei@hotmail.com
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Baseline Characteristics, Outcome Measures, Adverse Events and so on
Supporting Information: CSR
URL: https://www.medicalresearch.org.cn/login